CLINICAL TRIAL: NCT02664298
Title: Prospective Registry of Immediate/Delayed Loading of Implants in the Cranial Bone-grafted Severely Atrophic Jaw
Acronym: ILICRAN
Status: Terminated | Type: Observational
Why Stopped: Registry of patients registry has been discontinued
Sponsor: AZ Sint-Jan AV (Other)
Responsible Party: Principal Investigator, Johan Abeloos, Maxillofacial Surgeon, Head of Department, AZ Sint-Jan AV
Other Study IDs: B049201525497
Record Dates: First submitted 2016-01-11; First posted 2016-01-27 (Estimated); Last update posted 2022-02-28 (Actual); Status verified 2022-02

CONDITIONS: Jaw, Edentulous; Jaw, Partially Edentulous
Keywords: severely atrophic jaw; cranial bone-graft; dental implants; immediate loading; augmentation maxilla/mandible; sinus-floor elevation/sinuslift; dental prosthesis; implant supported; provisional implants; temporary implants; one-stage surgery; alveolar ridge augmentation; maxilla
MeSH Terms: conditions — Jaw, Edentulous; Jaw, Edentulous, Partially

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 36 Months
Oversight: Data Monitoring Committee: No

SUMMARY:
Edentulism is often associated with a negative psychosocial impact. The concept of prosthetic rehabilitation in which a prosthesis is supported by osseointegrated implants, was first introduced in the late 1960s by Brånemark et al. and offers an interesting alternative to removable prosthesis. However, for patients with a severely atrophic maxilla or mandible, cranial bone grafting of the jaw is required to increase bone width and height necessary for implant insertion. An active collaboration between the surgeons from the Oral and Maxillofacial Department and the prosthodontist from the Department of Dentistry has been established for continuous quality improvement of the concept of (immediate/delayed) implant loading in patients requiring cranial bone grafts to augment their severely atrophic jawbone.

The investigators aim to develop a prospective database registering (immediate/delayed) implant loading data of all patients eligible according to the protocol. Patient demographics, surgical, dental, prosthetic and patient satisfaction parameters are collected during consecutive visits within the framework of routine practice.

Development of a database registering immediate functional loading data secondary to cranial bone-grafting of a severely atrophic jaw, will provide more information about potential patient, surgical and prosthetic factors influencing long-term biological and mechanical stability, as well as patient satisfaction. Moreover, registration of those results could function as a measurement of quality of care, and could be used for sample size calculation for future large prospective trials.

ELIGIBILITY:
Inclusion Criteria:

* Patients of all ages
* Patients of all genders
* Patients with moderate to extreme bone atrophy of the jaw (class IV to VI according to Cawood and Howell (Cawood & Howell, 1988), caused by terminal periodontitis or edentulism
* Patients requiring bone augmentation procedures through cranial bone grafting for jaw reconstruction
* Patients ineligible for conventional removable prosthetic rehabilitation

Exclusion Criteria:

* Patients not eligible according to abovementioned criteria
* Patients with severe uncontrolled diabetes
* Patients with cranial vault without diploe and/or cranial vault thickness <3mm, as defined with cone-beam CT (De Ceulaer, et al., 2012)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: all consenting patients that require fixed prosthetic rehabilitation in a cranial bone-grafted severely atrophic jaw
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2007-01 (Actual); Primary Completion 2021-02 (Actual); Study Completion 2021-02 (Actual)

PRIMARY OUTCOMES:
IPI survival rate at time of immediate loading in patients with cranial bone-grafted severely atrophic jaw | within 6 months postsurgery
definitive implant survival rate in patients with cranial bone-grafted severely atrophic jaw | within 12 months postoperative
bone-graft resorption, as evaluated through cone-beam computed tomography | within 12 months postoperative
prosthesis survival rate | until a maximum of 10 years follow-up
bone-graft resorption, as evaluated through cone-beam computed tomography | until a maximum of 10 years follow-up

SECONDARY OUTCOMES:
Prevalence of patients with severely atrophic jaw requiring cranial bone-grafting | every 12 months, until a maximum of ten years
Potential biologic or mechanical risk factors that could predict undesirable functional or aesthetic outcome, through regression analysis | within 12 months postsurgery

OTHER OUTCOMES:
patient satisfaction, through visual analogue scale | within 12 months postsurgery (short-term); at annual follow-up until a maximum of 10 years follow-up (long-term)

CONTACTS AND LOCATIONS:
Overall Officials: Johan Abeloos, MD, Principal Investigator — Department of Oral and Maxillofacial Surgery, General Hospital Saint-John Bruges, Bruges, Belgium
Locations (1):
- Araceli Diez-Fraile, Bruges, Other (Non U.s.), Belgium

IPD SHARING:
Plan to Share IPD: No